CLINICAL TRIAL: NCT05412316
Title: Test-Retest Reliability of an Experimental Model of Shoulder Muscle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Leonardo Intelangelo, Head of the University Center for Assistance, Teaching and Research, University of Gran Rosario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: approval number 04/22
Record Dates: First submitted 2022-05-31; First posted 2022-06-09 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Musculoskeletal Pain
Keywords: Short-wave diathermy; Experimental pain model; Muscle pain; Generalized hypersensitivity; Shoulder pain
MeSH Terms: conditions — Musculoskeletal Pain; Myalgia; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: The SWD will be applied using a CEC M-8 shortwave thermotherapy unit (CEC Electrónica S.R.L., Argentina) that emits RF at a frequency of 27.12 MHz. The device has two rectangular capacitive applicators (18 × 12 cm), which will be placed below and above the dominant shoulder. The coplanar application will be done using the continuous wave mode. The intensity of SWD will be gradually increased until the volunteer perceives a sensation of heat, and once familiar with this perception, the intensity will be increased until a sensation of constant but tolerable pain is evoked. This sensation will be maintained throughout the SWD application. Once the first application is completed, the volunteer will be allowed to rest for a period of 2-3 minutes and three repetitions will be performed. Healthy volunteers will be in a lateral supine position, and a cotton towel will be used to absorb perspiration and avoid unwanted heat effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Healthy volunteers that fulfill the inclusion criteria. Intervention: Short-wave diathermy (Radiation)
  Interventions: Other: Intervention: Short-wave diathermy

INTERVENTIONS:
Other: Intervention: Short-wave diathermy — The SWD will be applied using a CEC M-8 shortwave thermotherapy unit (CEC Electrónica S.R.L., Argentina) that emits RF at a frequency of 27.12 MHz. The device has two rectangular capacitive applicators (18 × 12 cm), which will be placed below and above the dominant shoulder. The coplanar application will be done using the continuous wave mode. The intensity of SWD will be gradually increased until the volunteer perceives a sensation of heat, and once familiar with this perception, the intensity will be increased until a sensation of constant but tolerable pain is evoked. This sensation will be maintained throughout the SWD application, and three repetitions will be performed. Healthy volunteers will be in a lateral supine position, and a cotton towel will be used to absorb perspiration and avoid unwanted heat effects.

SUMMARY:
High frequency oscillations of non-ionizing electromagnetic fields range can heat deep tissues in a well-localized region. Recently, a new SWD-based model showed to be a promising tool for investigating muscle pain in humans. The main advantages of the model are its noninvasiveness, the ability to control stimulation parameters, and the convenience of the time frame in which pain and hyperalgesia are developed. This study assess the reliability of SWD pain model to induced transient and intensity-controlled muscle soreness on shoulder in healthy volunteers.

DETAILED DESCRIPTION:
This Test-Retest Reliability study comprises a sample of 31 healthy volunteers. Volunteers will be invited to participate in the study through social networks and e-mail.

Experimental pain model assessment

The radiofrequency electromagnetic fields can be produced in the range of 3 kHz to 300 GHz, but frequencies around 27 MHz (short-wave) are preferred to heat deep tissues. Deep tissue heating by means of RF is a safe and extensively used technique in palliative treatment of pain and as a healing agent in soft tissues. This study assess the reliability of SWD to induce soreness. The study will be conducted in two experimental sessions on different days, at least 48 to 72 hours apart each other in order to avoid carryover effects. In each experimental session, several measures will be performed to assess different physiological parameters, including: pressure pain thresholds (PPT), specific self-report questionnaire, isometric muscle strength, pain distribution and myoelectric activity.

In the first session (Test), participants will be interviewed to collect anthropometric data and health history. Basic upper quadrant physical examination will be performed to check inclusion and exclusion criteria. Before and after the application of SWD, several assessments will be performed. Among the different assessment, myoelectric activity of infraspinatus and deltoid muscle will be recorded during isometric arm lifting task. The isometric task will consist in maintaining the arm in 90 degree elevation in the scapular plane (arm flexion) for 8 seconds. This task will be repeated 5 times with 15 seconds of rest between each trial. Finally, a fatiguing motor task will be performed, consisting of flexion and extension of the arm executed cyclically in a range of motion between 30 and 90 degree in the scapular plane. To ensure fatigue, volunteers will perform the task with an additional weight. The size of the weight will be calculated according to each volunteer body mass (1.25 kg in participants under 68 kg and 2.5 kg in participants over 68 kg). The arm flexion and extension speed will be guided using a 60 beats/s metronome. Same process will be repeated in the second session (Retest).

Sample size considerations:

All the reliability assessment methods used in this study are related to the within-subject standard deviation (SD_w). For a test-retest experiment, the SD_w can be calculated as〖 SD〗_w=(SD_diff)⁄√2, and the LoA can be reformulated as bias ± 1.96 〖SD〗_w √2. The precision to estimate SD_w depends on both the number of subjects, n, and the number of observations per subject. A sample size of 31 subjects is required considering a confidence interval of 25% at either side of the estimation of SD_w, and for m=2 observations per subject.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the content and scope of the experiment, and compliance with the experiment's instructions.
* To have signed the informed consent.

Exclusion Criteria:

* Pregnancy.
* Previous history of neurological or musculoskeletal disorders or chronic pain.
* Previous history of addictive behavior, defined as abuse of alcohol, cannabis, opioids or other drugs.
* Previous history of thermosensitivity disorders.
* Previous history of mental illness.
* Presence of fever, tuberculosis, tumors, infectious processes, or acute inflammatory processes.
* Implantation of peacemaker or metallic prosthesis.
* Use of analgesics within 24 h prior to the experiment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) | At baseline and 30 - 60 minutes after of SWD.
  Change in the PPT (kPa) will be assessed bilaterally over the medial portion of the infraspinatus muscle using a digital algometer (Somedic SenseLab AB, Sweden) with a 1-cm2 round tip. Pressure will be gradually increased from 0 kPa at a rate of approximately 50 kPa/s (maximal achievable pressure: 2,000 kPa). The volunteers will be asked to press the button when they perceive that the pressure changes to pain, stopping the estimation at this point. The assessment will be repeated 3 times for each sides, alternating sides between measurements. Each measure will be performed at 30-second intervals.

SECONDARY OUTCOMES:
Pain distribution | At 30 - 60 minutes after the application of SWD.
  Extension of the reported pain drawings. The results will be expressed as the percentage of the total body area.
Modified Likert scale | At 30 - 60 minutes after the application of SWD.
  A modified self-report Likert scale was used to follow the temporal progression of muscle pain/soreness after SWD, with 0 defining a complete absence of soreness and 6 indicating severe soreness.
Myoelectrical activity (EMG) | At 10 minutes before and 30 - 60 minutes after the application of SWD.
  Change in muscle activity will be assessed. Monopolar multichannel recording (6 channels) will be distributed spatially across the infraspinatus muscle, and monopolar channels will be recorded for the medial and posterior deltoid muscle. BIOAMP Biopotential amplifier will be used for recording the EMG signals, 8-channel (sample rate: 2 KHz) (UNER, Argentina) during execution of the motor tasks. EMG will be recorded before and 30 - 60 minutes after SWD application to assess redistribution of the muscle activity induced by the transient pain.
Isometric muscle strength | At baseline and 30 - 60 minutes after the application of SWD.
  Change in the maximal isometric strength (kgf) for external rotation in dominant shoulder will be assessed using a Hand Held Dynamometer (Lafayette Manual Muscle Testing System, Model 01165, Lafayette, IN). The measures will be taken with the volunteers in the standing position, and the arm will be placed at the side of the body with the elbow flexed at 90º, and the forearm in neutral pronosupination. The examiner will be held the dynamometer at the dorsal aspect of the distal third of the forearm. Three 6-seconds measures will be taken with rest between them and the peak and mean value will be calculated.
Visual analog scale | During the application of SWD.
  A continuous visual analog scale ranging from 0 to 100, where 0 represents no perception, 30 represents pain threshold (defined as the time to reach a painful sensation at the predefined stimulation intensity) and 100 represents the tolerance threshold (defined as the sensation of pain when becomes intolerable)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gran Rosario, Rosario, Santa Fe Province, Argentina

REFERENCES:
- [Background] Biurrun Manresa JA, Fritsche R, Vuilleumier PH, Oehler C, Morch CD, Arendt-Nielsen L, Andersen OK, Curatolo M. Is the conditioned pain modulation paradigm reliable? A test-retest assessment using the nociceptive withdrawal reflex. PLoS One. 2014 Jun 20;9(6):e100241. doi: 10.1371/journal.pone.0100241. eCollection 2014. PMID 24950186